CLINICAL TRIAL: NCT02304926
Title: Study of Lipoprotein Subfractions, Inflammation, Oxidative Stress and Endothelial Function After Treatment With Simvastatin and Ezetimibe Administered Alone and in Combination in Hyperlipidemic Patients
Brief Title: Effects of Simvastatin and Ezetimibe on Cardiovascular Risk Markers in Patients With Dyslipidemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Antonio Hernandez Mijares, MD, Phd, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIM-EZE-2009-01
Record Dates: First submitted 2014-11-25; First posted 2014-12-02 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: Dyslipidemia
Keywords: Dyslipidemia; Simvastatin; Ezetimibe; Lipid profile; Inflammation; Oxidative stress; Endothelial function
MeSH Terms: conditions — Dyslipidemias; Inflammation | interventions — Simvastatin; Ezetimibe; Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin (Experimental): Hyperlipidemic patients received simvastatin (40 mg/day) for 4 weeks, after they were administered combined therapy (simvastatin, 40 mg/day plus ezetimibe,10 mg/day) for an additional 4-week period. Lipid profile, lipoprotein subfractions of LDL and HDL, inflammatory, oxidative stress and endothelial function parameters were evaluated.
  Interventions: Drug: Simvastatin; Drug: Simvastatin + Ezetimibe
- Ezetimibe (Experimental): Hyperlipidemic patients received ezetimibe (10 mg/day) for 4 weeks, after they were administered combined therapy (simvastatin, 40 mg/day plus ezetimibe,10 mg/day) for an additional 4-week period. Lipid profile, lipoprotein subfractions of LDL and HDL, inflammatory, oxidative stress and endothelial function parameters were evaluated.
  Interventions: Drug: Ezetimibe; Drug: Simvastatin + Ezetimibe

INTERVENTIONS:
Drug: Simvastatin — simvastatin (40 mg/day) for 4 weeks
  Arms: Simvastatin
Drug: Ezetimibe — ezetimibe (10 mg/day) for 4 weeks
  Arms: Ezetimibe
Drug: Simvastatin + Ezetimibe — combined therapy simvastatin (40 mg/day) + ezetimibe (10 mg/day) for 4-week period

SUMMARY:
Coadministration of drugs is common in the pharmacologic treatment of dyslipidemia, with statins and ezetimibe generally constituting the medication of choice. By acting at different levels, the combination of these drugs allows the therapeutic objective to be achieved. However, it is not known how these drugs qualitatively affect the composition of lipoprotein subfractions, which differ in size and atherogenic potential. The investigators set out to evaluate this effect as well as their effects on inflammatory, oxidative stress and endothelial function parameters.

DETAILED DESCRIPTION:
The study consisted of a randomised parallel trial and took place during a period of 2 months. A total of 42 hyperlipidemic patients were randomly assigned to one of 2 groups: one received simvastatin (40 mg/day) and the other received ezetimibe (10 mg/day) for 4 weeks, after which both groups were administered combined therapy for an additional 4-week period. Lipid profile, lipoprotein subfractions of LDL and HDL, inflammatory, oxidative stress and endothelial function parameters were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* LDL cholesterol concentration of between 160-190 mg/dl in patients with less than 2 cardiovascular risk factors
* LDL concentration of between 130-160 mg/dl in patients that presented 2 or more cardiovascular risk factors.

Cardiovascular risk factors were defined as: age (≥ 45 years in men and ≥55 years in women), a smoking habit, hypertension (≥140/90 mmHg), diabetes mellitus, a high-density lipoprotein (HDL) cholesterol concentration of ≤ 40mg/dl, and a family history of cardiovascular disease.

Exclusion Criteria:

* Triglyceride concentration > 400 mg/dl
* Diabetes Mellitus
* Kidney, liver, or thyroid disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hernández, MD, Phd, Principal Investigator — FISABIO - University Hospital Dr Peset

REFERENCES:
- [Background] Berneis K, Rizzo M, Berthold HK, Spinas GA, Krone W, Gouni-Berthold I. Ezetimibe alone or in combination with simvastatin increases small dense low-density lipoproteins in healthy men: a randomized trial. Eur Heart J. 2010 Jul;31(13):1633-9. doi: 10.1093/eurheartj/ehq181. Epub 2010 Jun 6. PMID 20525999
- [Background] Florentin M, Liberopoulos EN, Moutzouri E, Rizos CV, Tselepis AD, Elisaf MS. The effect of simvastatin alone versus simvastatin plus ezetimibe on the concentration of small dense low-density lipoprotein cholesterol in subjects with primary hypercholesterolemia. Curr Med Res Opin. 2011 Mar;27(3):685-92. doi: 10.1185/03007995.2010.546394. Epub 2011 Jan 27. PMID 21271793
- [Background] Bays HE, Ose L, Fraser N, Tribble DL, Quinto K, Reyes R, Johnson-Levonas AO, Sapre A, Donahue SR; Ezetimibe Study Group. A multicenter, randomized, double-blind, placebo-controlled, factorial design study to evaluate the lipid-altering efficacy and safety profile of the ezetimibe/simvastatin tablet compared with ezetimibe and simvastatin monotherapy in patients with primary hypercholesterolemia. Clin Ther. 2004 Nov;26(11):1758-73. doi: 10.1016/j.clinthera.2004.11.016. PMID 15639688

RESULTS

PARTICIPANT FLOW:
Groups:
- Simvastatin: 20 hyperlipidemic patients received simvastatin (40 mg/day) for 4 weeks, after they were administered combined therapy (simvastatin, 40 mg/day plus ezetimibe,10 mg/day) for an additional 4-week period. Lipid profile, lipoprotein subfractions of LDL and HDL, inflammatory, oxidative stress and endothelial function parameters were evaluated.
  Simvastatin: simvastatin (40 mg/day) for 4 weeks
  Simvastatin + Ezetimibe: combined therapy simvastatin (40 mg/day) + ezetimibe (10 mg/day) for 4-week period
- Ezetimibe: 20 hyperlipidemic patients received ezetimibe (10 mg/day) for 4 weeks, after they were administered combined therapy (simvastatin, 40 mg/day plus ezetimibe,10 mg/day) for an additional 4-week period. Lipid profile, lipoprotein subfractions of LDL and HDL, inflammatory, oxidative stress and endothelial function parameters were evaluated.
  Ezetimibe: ezetimibe (10 mg/day) for 4 weeks
  Simvastatin + Ezetimibe: combined therapy simvastatin (40 mg/day) + ezetimibe (10 mg/day) for 4-week period
Period: Overall Study
Arm/Group | Simvastatin | Ezetimibe
Started | 22 | 20
Completed | 20 | 19
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin | Ezetimibe | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (12.7) | 57.6 (10.2) | 57.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 5 | 3 | 8
Body mass index [Mean (Standard Deviation); unit: Kg/m2] | 28.6 (3.9) | 31.2 (7.3) | 29.8 (5.6)
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 133 (17) | 137 (14) | 134 (15)
Diastolic blood pressure (mm Hg) [Mean (Standard Deviation); unit: mm Hg] | 79 (10) | 80 (7) | 80 (8)

OUTCOME MEASURES:

1. Primary Outcome: Total Cholesterol Before and After Simvastatin/Ezetimibe Administration
Description: Total cholesterol concentration was measured by enzymatic assay
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
mg/dl
  Baseline | 255 (34) | 253 (26)
  4 weeks | 180 (29) | 215 (33)
  8 weeks | 173 (38) | 169 (39)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p < 0.05, ANOVA

2. Primary Outcome: Low-density Lipoprotein Cholesterol (LDLc) Before and After Simvastatin/Ezetimibe Administration
Description: Low-density lipoprotein cholesterol (LDLc) concentration was calculated using the method of Friedewald.
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
mg/dl
  Baseline | 178 (26) | 172 (29)
  4 weeks | 106 (18) | 138 (32)
  8 weeks | 98 (28) | 94 (36)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p < 0.05, ANOVA

3. Secondary Outcome: Levels of High-sensitive C-reactive Protein (hsCRP) Before and After Simvastatin/Ezetimibe Administration
Description: Levels of high-sensitive C-reactive protein (hsCRP) were analysed by a latex-enhanced inmunonephelometric assay
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: mg/l
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
mg/l
  Baseline | 4.02 (3.49) | 4.43 (4.97)
  4 weeks | 2.82 (2.69) | 3.98 (3.65)
  8 weeks | 2.64 (2.21) | 3.31 (3.48)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p < 0.05, ANOVA

4. Secondary Outcome: Levels of Interleukin-6 (IL-6) Before and After Simvastatin/Ezetimibe Administration
Description: Levels of proinflammatory cytokines (interleukin-6 (IL-6)) were analysed with a Luminex® 200™ system
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
pg/ml
  Baseline | 2.44 (1.62) | 2.94 (1.45)
  4 weeks | 2.83 (1.66) | 3.93 (2.28)
  8 weeks | 4.43 (4.30) | 5.78 (3.98)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p > 0.05, ANOVA

5. Secondary Outcome: Levels of Tumor Necrosis Factor α (TNF-α) Before and After Simvastatin/Ezetimibe Administration
Description: Levels of proinflammatory cytokines (tumor necrosis factor α (TNF-α)) were analysed with a Luminex® 200™ system
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
pg/ml
  Baseline | 3.43 (1.87) | 3.01 (2.29)
  4 weeks | 3.99 (1.77) | 5.09 (5.23)
  8 weeks | 4.43 (4.30) | 4.35 (4.09)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p > 0.05, ANOVA

6. Primary Outcome: High-density Lipoprotein Cholesterol (HDLc) Before and After Simvastatin/Ezetimibe Administration
Description: High-density lipoprotein cholesterol (HDLc) concentration was measured using a direct method
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
mg/dl
  Baseline | 47 (11) | 53 (15)
  4 weeks | 50 (13) | 53 (11)
  8 weeks | 51 (13) | 53 (13)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p < 0.05, ANOVA

7. Primary Outcome: Triglycerides Before and After Simvastatin/Ezetimibe Administration
Description: Triglyceride concentration were measured by enzymatic assay
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
mg/dl
  Baseline | 141 [104 to 168] | 120 [81 to 184]
  4 weeks | 117 [82 to 136] | 105 [81 to 142]
  8 weeks | 104 [82 to 146] | 81 [61 to 137]
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p < 0.05, ANOVA

8. Secondary Outcome: Mitochondrial Oxygen (O2) Consumption Before and After Simvastatin/Ezetimibe Administration
Description: Oxidative stress markers (mitochondrial oxygen (O2) consumption) was measured at baseline and after treatment by Clark electrode
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: Nmol O2/min/million cells
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
Nmol O2/min/million cells
  Baseline | 1.09 (0.15) | 1.09 (0.15)
  4 weeks | 1.54 (0.12) | 1.31 (0.13)
  8 weeks | 1.76 (0.21) | 1.67 (0.10)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p < 0.05, ANOVA

9. Secondary Outcome: Reactive Oxygen Species (ROS) Production Before and After Simvastatin/Ezetimibe Administration
Description: Oxidative stress markers (Reactive oxygen species (ROS) production) was measured at baseline and after treatment by fluorometric techniques
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: Fluorescence Units
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
Fluorescence Units
  Baseline | 74.7 (8.1) | 72.8 (8.3)
  4 weeks | 57.2 (8.9) | 63.5 (10.3)
  8 weeks | 43.3 (7.9) | 48.9 (3.3)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p < 0.05, ANOVA

10. Secondary Outcome: Membrane Potential Before and After Simvastatin/Ezetimibe Administration
Description: Oxidative stress markers (membrane potential) was measured at baseline and after treatment by fluorometric techniques
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: Fluorescence Units
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
Fluorescence Units
  Baseline | 46.6 (5.8) | 48.4 (3.9)
  4 weeks | 62.5 (5.4) | 56.7 (5.4)
  8 weeks | 70.4 (8.4) | 67.5 (4.5)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p < 0.05, ANOVA

11. Secondary Outcome: Levels of Glutathione (GSH) Before and After Simvastatin/Ezetimibe Administration
Description: Oxidative stress markers (levels of glutathione (GSH)) was measured at baseline and after treatment by fluorometric techniques
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: Fluorescence Units
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
Fluorescence Units
  Baseline | 2.68 (0.63) | 2.85 (0.71)
  4 weeks | 5.67 (0.59) | 3.79 (0.67)
  8 weeks | 7.92 (1.24) | 7.51 (1.09)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p < 0.05, ANOVA

12. Secondary Outcome: Leukocyte Rolling Flux Before and After Simvastatin/Ezetimibe Administration
Description: Interactions between leukocytes and human umbilical vein endothelial cells were evaluated by flow chamber microscopy. Leukocyte rolling was estimated as the number of leukocytes rolling over 100 μm2 of the endothelial monolayer during a 1-min period.
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: polymorphonuclear cells/min
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
polymorphonuclear cells/min
  Baseline | 412 (132) | 421 (203)
  4 weeks | 225 (61) | 392 (187)
  8 weeks | 147 (51) | 196 (99)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p < 0.05, ANOVA

13. Primary Outcome: Non-HDL Cholesterol Before and After Simvastatin/Ezetimibe Administration
Description: Non-HDLc concentration was obtained by calculating the difference between total cholesterol and HDLc
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
mg/dl
  Baseline | 208 (29) | 200 (28)
  4 weeks | 130 (23) | 162 (33)
  8 weeks | 122 (31) | 115 (39)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p < 0.05, ANOVA

14. Primary Outcome: Low Density Lipoprotein Size Before and After Simvastatin/Ezetimibe Administration
Description: LDL subfractions were separated by high-resolution polyacrylamide gel tubes using the Lipoprint® system. The LDL electrophoretic profile allows 2 patterns to be defined: pattern A or large and buoyant LDL, and pattern non-A or small and dense LDL.
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: Angström
Groups:
- Ezetimibe: 19 hyperlipidemic patients received ezetimibe (10 mg/day) for 4 weeks, after they were administered combined therapy (simvastatin, 40 mg/day plus ezetimibe,10 mg/day) for an additional 4-week period. Lipid profile, lipoprotein subfractions of LDL and HDL, inflammatory, oxidative stress and endothelial function parameters were evaluated.
  Ezetimibe: ezetimibe (10 mg/day) for 4 weeks
  Simvastatin + Ezetimibe: combined therapy simvastatin (40 mg/day) + ezetimibe (10 mg/day) for 4-week period
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
Angström
  Baseline | 268.1 (4.7) | 270.4 (2.3)
  4 weeks | 270.4 (2.9) | 271.5 (2.2)
  8 weeks | 271.7 (2.7) | 272.0 (1.9)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p < 0.05, ANOVA

15. Secondary Outcome: Leukocyte Adhesion Before and After Simvastatin/Ezetimibe Administration
Description: Interactions between leukocytes and human umbilical vein endothelial cells were evaluated by flow chamber microscopy. Adhesion was evaluated by counting the number of polymorphonuclear cells that maintained stable contact with human umbilical vein endothelial cells (HUVEC) for 30 seconds.
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: polymorphonuclear cells/mm2
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
polymorphonuclear cells/mm2
  Baseline | 25.1 (8.2) | 25.6 (12.1)
  4 weeks | 15.0 (4.1) | 23.8 (14.2)
  8 weeks | 10.9 (2.5) | 12.5 (4.9)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p < 0.05, ANOVA

16. Secondary Outcome: Leukocyte Rolling Velocity Before and After Simvastatin/Ezetimibe Administration
Description: Interactions between leukocytes and human umbilical vein endothelial cells were evaluated by flow chamber microscopy.The rolling velocity in the field of focus was determined by measuring the time required by 20 consecutive leukocytes to cover a distance of 100 μm.
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: micrometer/second
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
micrometer/second
  Baseline | 469 (53) | 524 (43)
  4 weeks | 553 (54) | 533 (42)
  8 weeks | 608 (43) | 629 (34)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p < 0.05, ANOVA

17. Primary Outcome: Apolipoprotein B Before and After Simvastatin/Ezetimibe Administration
Description: Levels of apolipoprotein B were determined by inmunonephelometry
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
mg/dl
  Baseline | 139 (20) | 127 (23)
  4 weeks | 92 (18) | 110 (24)
  8 weeks | 84 (18) | 79 (29)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p < 0.05, ANOVA

18. Secondary Outcome: Levels of Vascular Cell Adhesion Molecule 1 (VCAM-1) Before and After Simvastatin/Ezetimibe Administration
Description: The vascular cell adhesion molecule 1 (VCAM-1) was evaluated in serum by Luminex® 200™ system
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
ng/ml
  Baseline | 1314 (251) | 1371 (342)
  4 weeks | 1137 (407) | 1166 (526)
  8 weeks | 1074 (385) | 1220 (201)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p > 0.05, ANOVA

19. Secondary Outcome: Levels of Intercellular Adhesion Molecule 1 (ICAM-1) Before and After Simvastatin/Ezetimibe Administration
Description: The intercellular adhesion molecule 1 (ICAM-1) was evaluated in serum by Luminex® 200™ system
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
ng/ml
  Baseline | 188 (46.5) | 160.6 (37.8)
  4 weeks | 139.5 (53.4) | 114.7 (24.6)
  8 weeks | 122.2 (52.2) | 108.1 (36.1)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p < 0.05, ANOVA

20. Secondary Outcome: Levels of E-selectin Before and After Simvastatin/Ezetimibe Administration
Description: E-selectin was evaluated in serum by Luminex® 200™ system
Time Frame: Baseline, 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 20 | 19
ng/ml
  Baseline | 45.1 (21.0) | 39.7 (15.6)
  4 weeks | 38.9 (16.0) | 30.5 (14.7)
  8 weeks | 29.2 (11.0) | 24.4 (9.1)
Statistical Analysis 1: Comparison: Simvastatin vs Ezetimibe; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were not collected
Description: Adverse events were not collected
Groups:
- Adverse Events Were Not Collected; EG001: Adverse events were not collected
Arm/Group | Adverse Events Were Not Collected | EG001
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No